CLINICAL TRIAL: NCT01416701
Title: Vitamin D and COPD. A Randomised, Double-blind, Placebo-controlled Trial of the Effect of Vitamin D on Withdrawal From Pulmonary Rehabilitation and Exercise Endurance
Brief Title: Vitamin D and Chronic Obstructive Lung Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: It was not possible to enroll the planned amount of subjects. Many patients with chronic obstructive pulmonary disease already took large doses of vitamin D.
Sponsor: Jorgen Vestbo (Other)
Responsible Party: Sponsor-Investigator, Jorgen Vestbo, Prof. DMSc, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DvitKOL01022011
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Obstructive Lung Disease
Keywords: COPD; Vitamin D; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Vitamin D; Cholecalciferol; Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (D3, cholecalciferol) (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D (D3, cholecalciferol)
- Placebo (cellulose) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo (cellulose)

INTERVENTIONS:
Dietary Supplement: Vitamin D (D3, cholecalciferol) — Week 0-4: 152 mcg/daily (4 tablets) Week 5-52: 76 mcg/daily (2 tablets)
  Other Names: Bio Vinci Mega D-vitamin
  Arms: Vitamin D (D3, cholecalciferol)
Dietary Supplement: Placebo (cellulose) — Week 0-4: 4 tablets daily Week 4-52: 2 tablets daily
  Arms: Placebo (cellulose)

SUMMARY:
The purpose of this study is to examine the effect of vitamin D intervention in patients with chronic obstructive pulmonary disease (COPD) undergoing rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Diagnosed COPD with forced expiratory volume in 1 second (FEV1) < 50 % of predicted
* Breathlessness relative to MRC dyspnoea grade 3 or more

Exclusion Criteria:

* Patients with known diseases of bone metabolism apart from osteoporosis and patients with granulomatous disease
* Patients with hyper- or hypocalcemia at inclusion
* Patients with cardiovascular or musculoskeletal disease that impacts significantly on walking based on the investigator's judgement
* Patients with dementia or other mental conditions rendering them unable to understand the study information and thus provide informed consent
* Patients with terminal disease or known cancer with bone metastases, increasing their risk of hypercalcemia
* Patients taking more than 20 mcg vitamin D on a daily basis. If a patient takes vitamin D below this limit, dose should have been stable 6 months prior to inclusion in order to achieve steady-state.
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Withdrawal from rehabilitation. | 24 weeks
  Withdrawal will be defined as giving up rehabilitation or delaying any training visit by more than 3 weeks.
Improvement in walking distance | 24 weeks
  Change in walking distance from week 0 to week 24. Exercise capacity is evaluated using paced walking (Incremental Shuttle Walk Test(ISWT) and Endurance Shuttle Walk Test (ESWT)).

SECONDARY OUTCOMES:
Change in vitamin D status. | 52 weeks
  se-25-OHD se-PTH
Change in calcium metabolic status. | 52 weeks
  se-calcium se-phosphate se-magnesium
Change in quality of life. | 52 weeks
  COPD Assessment Test (CAT) and St George Respiratory Questionnaire (SGRQ).
Change in status of bone metabolism. | 52 weeks
  DXA (Dual energy X-ray Absorptiometry) scans
Change in walking distance. | 52 weeks
  Change in walking distance from week 0 to week 11 and week 52. Exercise capacity is evaluated using paced walking (Incremental Shuttle Walk Test (ISWT) and Endurance Shuttle Walk Test (ESWT)).
Change in fat mass and fat free mass. | 52 weeks
  Whole body DXA scans.
Change in physical activity. | 24 weeks
  Physical activity at home is measured over a week using an activity sensor (SenseWear Pro armband).
COPD exacerbations. | 52 weeks
All cause hospital admissions. | 52 weeks
All cause mortality. | 52 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Vestbo, DMSc, Principal Investigator — Hvidovre Universityl Hospital
Locations (2):
- Denmark (2):
  - Hvidovre University Hospital, Department of Respiratory Medicine, Hvidovre
  - Medical Unit, Hvidovre University Hospital, Hvidovre